# RADx-UP CDCC Rapid Research Pilot Program: "Culturally-relevant Community Connections (C3) to Increase COVID-19 Testing in the Black/African American Community"

Document Date: 02/22/2024

NCT05918952

## Purpose of the Study

The purpose of this study is to identify barriers and facilitators to COVID testing among members of the Black/African American community. The expected outcome of this project is to increase COVID testing among Black/African American community. The secondary aim is to examine the use of culturally relevant edutainment video messaging combined with trusted opinion leaders in the community as a strategy to increase COVID testing.

Aim 1. Provide testing to Black/African American communities throughout North Carolina through partnerships with beauty industry professionals in order to promote early detection of infected individuals and prevent asymptomatic and pre-symptomatic spread of COVID-19.

Aim 2. Develop and implement communication messages that will be disseminated in barbershops and beauty salons to examine the impact of culturally relevant messaging on uptake of COVID testing.

## **Background & Significance**

The pandemics of COVID-19 and racial discrimination in America have joined forces to illuminate inequalities in healthcare delivery and health outcomes of Black Americans. These pandemics have increased attention to the medical distrust, racism, discrimination, implicit bias, and unequal treatment that has occurred in this country for centuries.

Trusted venues such as barbershops and beauty salons are gatekeepers and facilitators of trusted information in the Black community. Our addressing Health disparities through Engagement, Equity, Advocacy, and Trust (HEEAT) Research Lab partners with barbers and stylists for health promotion in communities of color. We co-founded North Carolina Barbers and Stylists for Health Equity (NCBSHE), a network of barbershops and beauty salons serving primarily Black clientele throughout NC. NCBSHE is led by barbers and stylists, with academic partners serving the organization in non-leadership roles.

Due to barriers including access to care, discrimination, and medical distrust, engaging the Black community in health research and improvement activities requires a community-based approach. Our novel approach integrates evidence-based strategies that will address these barriers to engagement. Success of this project in increasing uptake of COVID-19 testing in the Black community will serve as a model for other health-related activities beyond COVID.

#### Research Approach

Our current and prior work1 addressing HIV prevention among Black women successfully trained stylists in the community to bring awareness and knowledge of pre-exposure prophylaxis (PrEP). The first three months of this COVID-19 project will focus on training stylists and barbers as Opinion Leaders (OLs), development of edutainment videos, and training of research staff. An NP will provide telehealth support to customers who test positive, and the Community Coordinator will facilitate the OL workshop. The workshop will include updates on COVID in the designated testing areas, CDC guidelines for COVID-19, clinical presentation, prevention strategies, testing, and telehealth policies and procedures, and roles and responsibilities of an OL. An OL serves as a community liaison between the researcher and the community. They do not serve as interventionists but are informed of research practices and current studies taking place in their community.

We will partner with an established communication strategist team we have previously worked with to co-develop culturally and socially relevant short clip edutainment videos.

OLs training as an evidence-based model to promote health. Without ready and convenient access to credible, peer-reviewed information, people in search of information about health and well-being appear to turn to trusted local information sources such as personal connections and trusted healthcare professionals. Kim and colleagues2 note the importance of social networks and local information sources among underserved communities. Training of beauty industry professionals as OLs has been promising. There is evidence that customer confidence is increased when stylists undertake workshops in preparation for sharing information.

Edutainment videos are an evidence-based intervention strategy for health promotion and prevention among communities of color. Grounded in transportation theory5, edutainment videos are designed to entertain and improve literacy while communicating prosocial norms and behaviors. These short clip videos will be accessible by scanning a QR code in the barbershop or beauty salon. A trained beauty professional will offer each client the opportunity to view the video. A \$5 off coupon for hair services with the designated salon/shop will be offered if the client watches the video. At the end of the video, the client will be asked if they would like to be tested that day. If they respond no, the client will be asked a set of questions that explain the reason (e.g., I was tested in the past 2-weeks, I prefer to get tested at my doctor's office, I don't think I have COVID, I don't trust the COVID test). If the customer says yes, the client will be asked a set of questions about the reason for the decision (facilitators) (e.g., I feel comfortable testing in this space, the video encouraged me to be tested today, I have been wanting to get tested, but did not have easy access to testing).

A nurse-led model of care: the role of the advanced practice nurse and telehealth. NPs are positioned to advance health equity and support efforts to improve testing in the community. In prior work by our team and others, the nursing workforce is increasingly being recognized as being uniquely positioned to drive healthcare innovation to advance health equity. A recent National Academies of Sciences, Engineering, and Medicine (NASEM) report outlined a comprehensive vision for nurse-led innovation as a driving force in overhauling conventional models of health service delivery. Specifically, the NASEM report endorses the scale-up of nurse-led interdisciplinary care delivered directly in community settings. The NP will be a liaison for OLs and salons/shops and will contact customers who test positive for COVID to educate them of next steps. Since COVID, telehealth has been used to improve access to care and address barriers such as transportation, childcare limitations, and needing time off for appointments.9 Telehealth addresses traditional barriers to and disparities in access to care while also improving efficiency.

## **Design & Procedures**

Participants will have access to a QR code via a flier located in the salon/barbershop. The QR code will take them to the screening and study information sheet for the participant to review. A link to the communications video will be embedded at the end of the study information sheet.

The communications video will also discuss components of the study information sheets, including the purpose of the study, and information regarding covid and proper covid testing procedures.

At the end of the video, the potential participant will be asked if they are interested in taking a covid test. Study information sheets will also be available in the private designated testing area for participants to review after watching the communications video.

All participants will be asked questions regarding their experience with the communications video, covid-19 testing decision-making process, and demographic data. This data will take approximately 10 minutes to complete. By completing demographic and survey questions you are agreeing to participate in this research study.

The participant will have access to the covid test in the private designated testing area.

All Participants (those who tested and those who did not) will receive a follow-up call within 3 months of consenting with an invitation to attend the community conversation centered around Black/African American health in the local community where they will be invited to complete the RADx-UP survey.

Participants who are not receiving services but are interested in participating can participate and will receive a gift bag that consists of water bottles and a journal (Value \$5).

The study team will participate in two community events whereby we will offer testing and outreach/education about COVID-19. The study team will provide gift bags for participants that consist of water bottles and a journal (Value \$5).

Hold focus group meetings with 10-12 people from each testing site. These will not be combined, and all participants will be customers of the OL's salon on shop. 4 focus groups will be held. Each participant in the focus group will be compensated with a \$50 Amazon gift card.

## Selection of Subjects

#### Eligibility Criteria

Customers (study participants) must self-identify, as Black or African American, be 18 or older, and visit the beauty salon or barber shop to enroll in the study.

**Subject Recruitment and Compensation** 

Two beauty salons and three barbershops have agreed to partner to implement this project. Recruitment of customers in these shops will take place through word of mouth, an IRB-approved recruitment flyer, and through the co-developed edutainment videos. On average, OL 1 in beauty salon 1 sees 40-60 customers per week; OL 2 in beauty salon 2 sees 30-50 clients per week; OL 3 in

barbershop 1 sees 60-100 customers per week; and OL 4 operates two barbershops seeing on average 200 customers per week.

The videos will give an overview and discuss the purpose of the study and will access to a link to the study information sheet. Study information sheets and study fliers will also be available in the salon and private designated testing area.

A \$5 off coupon for hair services with the designated salon/shop will be offered if the client watches the video. Coupons will be located in the private testing area.

## **Study Interventions**

Short clip videos being designed to discuss the testing process, the importance of getting tested and accessing care, and how COVID-19 has disproportionately affected the Black/African-American community.

#### **COVID Testing**

We propose to use the iHealth® Rapid COVID-19 Antigen Rapid Test. Per the EUA guidance, study participants will complete one test at a study location and receive one test to take home with instructions to complete it within 48 hours.

The first three months of this COVID-19 project will focus on training stylists and barbers as Opinion Leaders (OLs), development of edutainment videos, and training of research staff. An NP will provide telehealth support to customers who test positive, and the Community Coordinator will facilitate the OL workshop. Training will include updates on COVID in the designated testing areas, CDC guidelines for COVID-19, clinical presentation, prevention strategies, testing and telehealth policies, and procedures, and roles and responsibilities of an OL. OLs serve as a community liaison who has learned about the research process and current studies that involve their community.

There is evidence that customer confidence is increased when stylists undertake opinion leader workshop training in preparation for sharing information. This strategy focuses on building trust between the community and the research. Stylists will not serve as interventionists.

Each testing site will have a private designated space for customers to self-collect and test themselves privately. The edutainment video will serve as a resource for information on accurate test performance. Test one will be done in a private setting and results entered into REDcap and will also be written on a testing card with contact information for the purpose of follow-up. For test number two the customer will self-collect within 48 hours (per the FDA EUA for this particular test) and results will be entered into RedCap.

A locked box will be placed at the private designated testing area for customers who test, to put the card in. A QR code will be made available and accessible in the testing space that will take the participant to the study's REDCAP for them to enter their test results. They will also be provided with contact information for the NP (Dr. Ragan Johnson) if the customer tests positive. They will be available during business hours Monday through Friday. The Research Coordinator (Maralis Mercado Emerson) hired on this project will follow up with participants about testing two results. The RC will provide

contact information to the NP if the customer tests positive. Research Coordinator will collect testing cards on a bi-weekly basis.

Once contact has been made with the participant, the testing card will be disposed of in the provided sensitive shred. The research team has access to one in the IPE bldg. room 4232.

Risk/Benefit Assessment

Risks

No risks have been identified outside of the risk associated with self-testing

False Negatives:

To address potential false negatives, participants will take another test within 48 hrs. All test boxes will have the project QR code to the RedCap where participants will be able to provide test result information.

Risk may be involved with this study in the possibility that interview questions may be considered sensitive. Participants may refuse to answer any of the questions or stop study participation at any time. There is also the potential risk of loss of confidentiality. Every effort will be made to keep the information confidential; participants may use aliases.

Benefits

Participants will be contributing to best practices for engagement with potential future outbreaks.

## Data Analysis & Statistical Considerations

We anticipate 1000 study participants (200 per shop) based on the average number of clients who visit the salon/barbershop and the experience of the research team in recruiting and retaining this population for previous community engaged projects. Eligible subjects will include both participants who decide to get COVID testing as well as those who do not. We anticipate that estimated time to target accrual of 1000 will be April- October 2023. The NIH RADx-UP CDEs provide a standard set of study questions that RADx-UP projects are required to use in their COVID-19 testing studies. We will use data set from Tier 1 for this project. [176 items] Descriptive analysis will be used to summarize survey data and identify patterns from the specified data sample.

Demographic data will be collected from all participants to include sociodemographic Data, Housing employment and insurance, Work PPE and distancing, medical history, health status, disability, vaccine acceptance, testing, symptoms, alcohol and tobacco, and identity. Demographic information will summarized by mean and standard deviation for continuous variables and frequency and percentage for categorical variables.